CLINICAL TRIAL: NCT00753987
Title: Tolerability of Hypertonic Saline in Infants With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000008380
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Hypertonic Saline; Infants
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolerability of 7% hypertonic saline (Experimental): Administration of a single dose of 7% hypertonic saline
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: Hypertonic Saline — 5 ml of 7% saline will be administered via mask with Pari LC Plus nebuliser and a Pari Ultra Ned compressor.

SUMMARY:
The objective of the study is to determine whether or not inhalation of hypertonic saline will be tolerated by infants with cystic fibrosis and the effect of inhalation on their lung function.

DETAILED DESCRIPTION:
Cystic fibrosis lung disease is characterized by mucous retention which favors secondary bacterial infection and inflammation, which leads to lung damage and ultimately respiratory failure. Classically, therapeutic interventions are aimed to improve mucociliary clearance, to reduce both bacterial load and lower airway inflammation.

Hypertonic saline (HS) has been used for the induction of sputum production in all age groups to obtain secretions from the lower respiratory for diagnostic purposes. Hypertonic saline is also used in older children with CF, who do not produce sputum spontaneously, to obtain representative samples for microbiology.

There is evidence from studies in patients with cystic fibrosis that HS can improve mucociliary clearance. The improvement was more impressive in areas that were well ventilated, making it likely that HS will work better in patients with relatively preserved pulmonary function. Newer evidence also suggests that the osmotic effect on the airway surface that was expected to be short lived, may actually persist for longer time periods (up to 8 hours). All these data indicate that HS may be a useful agent in the treatment of CF patients.

As the effect on mucociliary clearance was found to be better in areas with adequate ventilation, it is logical to assume that treatment with HS may be most efficacious when initiated early in the disease process. So far, no data on the tolerability of inhalation of HS are available for infants with cystic fibrosis. However, evidence from infants with AIDS as well as recent studies in infants with bronchiolitis suggest that hypertonic saline can be safely administered by inhalation in infants. Nevertheless, proof of tolerability in CF infants is a prerequisite for longer term studies of HS in this age group. In older children, tolerability has been tested by measuring pulmonary function both before and after inhalation of HS saline. Similar data are not yet available for infants.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis
* Age 2 months to 2 years
* Routinely scheduled infant pulmonary function test.
* Clinical stability (no respirator tract infection for 4 weeks prior to study

Exclusion Criteria:

* Acute respiratory symptoms
* Wheezing at the time of study
* Supplemental oxygen therapy
* Oxygen saturation < 95 % on room air

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, FRCP(C), Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Interventional Trial: Hypertonic Saline: 5 ml of 7% saline will be administered via mask with Pari LC Plus nebuliser and a Pari Ultra Ned compressor.
Period: Overall Study
Arm/Group | Single Arm Interventional Trial
Started (13 were recruited) | 13 (13 participants were enrolled and 13 completed the studycompleted)
Completed (All 13 completed the study) | 13 (13 completed the study)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: infants with CF
Groups:
- Single Arm Study: Hypertonic Saline: 5 ml of 7% saline will be administered via mask with Pari LC Plus nebuliser and a Pari Ultra Ned compressor.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 13
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Age, continuous | 80.7 (31.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 13

OUTCOME MEASURES:

1. Primary Outcome: Decrease in FEV0.5 After Inhalation of Hypertonic Saline
Description: Number of participants with a decrease in FEV0.5 by 0% or more after inhalation of hypertonic saline. The number of participants with a change in FEV0.5 of *more than* 0% is reported.
Time Frame: 100 minutes
Population: 2 infants had to excluded, since they woke up before administration of the study medication and thus lung function measurements after administration could not be performed
Measure: Number; unit: participants
Groups:
- Decrease in FEV05: There was no decrease in lung function observed in the study in any subject
Arm/Group | Decrease in FEV05
Number analyzed (Participants) | 11
participants | 0

2. Secondary Outcome: Oxygen Saturation Below 92%
Description: Reduction of oxygen saturation below 92 % 10 minutes after inhalation of hypertonic saline. This change would be considered to reflect an abnormally low oxygen concentration and could reflect a negative impact of inhalation
Time Frame: 10 minutes
Measure: Number; unit: participants
Groups:
- Decrease in FEV05: Decrease in lung function measured by FEV 0.5 by more than 10 % after inhalation of hypertonic saline
Arm/Group | Decrease in FEV05
Number analyzed (Participants) | 11
participants | 0

3. Other Pre Specified Outcome: Number of Participants With Newly Detected Bacterial Pathogens on Throat Swab After Hypertonic Saline Inhalation
Description: Diagnostic yield of a throat swab for microbiological diagnosis of bacteria as measured by the number of participants with newly detected bacterial pathogens on respiratory culture after inhalation of hypertonic saline compared to previously performed throat swabs at the last clinic visit
Time Frame: 10 minutes after completion of inhalation
Population: CF infants
Measure: Number; unit: participants
Groups:
- Changes in Culture Positivity: within group comparison
Arm/Group | Changes in Culture Positivity
Number analyzed (Participants) | 13
participants | 0

4. Other Pre Specified Outcome: Number of Participants With Wheezing After Inhalation of Hypertonic Saline
Description: audible wheezing on auscultation 15 minutes after administration
Time Frame: 15 minutes
Population: Individuals with lung function data after inhalation
Measure: Number; unit: percentage of participants
Groups:
- Decrease in FEV05: There was no decrease in lung function observed in the study
Arm/Group | Decrease in FEV05
Number analyzed (Participants) | 11
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: throughout the test (2 hours)
Groups:
- SIngle Arm Trial: Hypertonic Saline: 5 ml of 7% saline will be administered via mask with Pari LC Plus nebuliser and a Pari Ultra Ned compressor.
Arm/Group | SIngle Arm Trial
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No